CLINICAL TRIAL: NCT00885391
Title: QT Variability Pre & Post Cardioversion in Patient's With Atrial Fibrillation
Brief Title: QT Variability Pre and Post Cardioversion
Acronym: DCCV
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Dawood Darbar, Associate Professor of Medicine and Pharmacology, Vanderbilt University
Other Study IDs: 060908; R01HL085690-01A2 (NIH)
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Cardioversion; Direct Current Cardioversion; QT Interval
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn whether the chemicals in the blood and urine are different when the heart is atrial fibrillation compared to normal sinus rhythm.

DETAILED DESCRIPTION:
Atrial Fibrillation variably activates the renin-angiotensin-aldosterone system (RAAS), stimulates the sympathetic nervous system, generates oxidant stress, produces natriuretic peptides, and increases ventricular rate. These are interrelated responses and the extent to which these or other pathophysiologic responses determine QT interval during and after Atrial Fibrillation (AF) is unknown. In this study, the QT variability is related to those potential markers in patients with AF undergoing elective DC-cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Scheduled to undergo an elective DC-Cardioversion of atrial fibrillation or atrial flutter at Vanderbilt University Medical Center

Exclusion Criteria:

* Undergoing emergent DC-Cardioversion of atrial fibrillation for hemodynamic instability
* Undergoing DC-Cardioversion for post-cardiac surgery
* Dual chamber pacemakers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology Clinic Hospital inpatient
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2007-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
QT variability before and after direct current cardioversion | 1.5

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Darbar, M.D., Ph.D., F.A.C.C., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States